CLINICAL TRIAL: NCT00585845
Title: A Phase 1, Open-Label, Dose-Escalation, Multiple Dose Study of the Safety, Tolerability, and Immune Response of CRS-207 in Adult Subjects With Selected Advanced Solid Tumors Who Have Failed or Who Are Not Candidates for Standard Treatment
Brief Title: Study of Safety and Tolerability of Intravenous CRS-207 in Adults With Selected Advanced Solid Tumors Who Have Failed or Who Are Not Candidates for Standard Treatment
Status: Terminated | Phase: Phase 1 | Type: Interventional
Sponsor: Anza Therapeutics, Inc. (Industry)
Responsible Party: Dung Thai, Anza Therapeutics, Inc.
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VAC07001
Record Dates: First submitted 2007-12-22; First posted 2008-01-03 (Estimated); Last update posted 2009-02-20 (Estimated); Status verified 2009-02

CONDITIONS: Malignant Epithelial Mesothelioma; Adenocarcinoma of the Pancreas; Carcinoma, Non-Small-Cell Lung; Adenocarcinoma of the Ovaries
Keywords: Cancer; Ovarian cancer; Pancreatic cancer; Non-small cell lung cancer; Mesothelioma; Mesothelin; Immunotherapy
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Neoplasms; Ovarian Neoplasms; Pancreatic Neoplasms; Mesothelioma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- CRS-207 (Experimental)
  Interventions: Biological: CRS-207, Live-attenuated Listeria monocytogenes expressing human Mesothelin

INTERVENTIONS:
Biological: CRS-207, Live-attenuated Listeria monocytogenes expressing human Mesothelin — 2-hour IV infusion once every 21 days, up to 4 doses. Doses from 1x10^8 cfu to 1x10^10 cfu.

SUMMARY:
This clinical trial will evaluate the safety and tolerability of CRS 207 an investigational product that is a weakened form (attenuated) of Listeria monocytogenes, a type of bacteria that is commonly found in the environment. CRS-207 has been altered in the lab to reduce its ability to cause disease, while maintaining stimulation of the immune system. CRS 207 has also been genetically modified with recombinant DNA to release an antigen called Mesothelin. Because CRS 207 stimulates an immune response to Mesothelin and Mesothelin may be present at higher levels on tumor cells than on normal cells, this clinical trial will also examine if CRS 207 boosts the immune system in a way that targets certain types of cancer.

The purpose of this first clinical trial with CRS-207 is to identify an appropriate dose of the investigation agent for later clinical studies and to explore safety when given to consenting adults with advanced cancer of the ovary or pancreas, non-small cell lung cancer, or advanced malignant epithelial mesothelioma. Immunological response to CRS-207 and tumor status of study participants will also be measured. Patients who choose to enter the study must meet all study entry criteria and must have previously failed standard treatment for their cancer. Qualifying study patients will be assigned to receive one of several dose levels of CRS-207. Each patient may receive up to 4 intravenous administrations (21 days apart) of CRS-207 at their assigned dose level.

DETAILED DESCRIPTION:
Patients who consent to participate in the study will be evaluated for eligibility according to their medical history, physical examination, blood testing, and computed tomography (CT) scan of thorax, abdomen, and pelvis. Those patients who qualify for the study will receive up to 4 intravenous doses of CRS-207, 21 days apart. After each infusion, they will be monitored overnight in an in-patient facility, including collection of blood specimens. Study participants will return after each infusion for outpatient follow-up visits for further blood tests and additional monitoring of safety and immune response to CRS-207. Participants will have repeat CT scans to measure tumor size after the 2nd dose and again after the 4th dose. On Day 91 participants will be discharged from the study. All study participants will be eligible to participate in a long-term follow-up study with a visit 6 months after the final dose of CRS-207 and annually thereafter for evaluation of disease progression, survival, and potential long-term toxicity of CRS 207.

ELIGIBILITY:
Inclusion Criteria:

1. Documented malignant epithelial mesothelioma, cancer of the pancreas or ovaries or non-small-cell lung cancer (NSCLC) and who have failed (or are not candidates for) standard therapy
2. ECOG Performance Status of 0 to 1, or Karnofsky Performance Status (KPS) of 80-100%
3. Adequate organ function as defined by study-specified laboratory tests
4. Must use acceptable form of birth control through the study and for 28 days after final dose of study drug
5. Signed informed consent form
6. Willing and able to comply with study procedures

Exclusion Criteria:

1. History of infection with Listeria, prior vaccination with a listeria-based vaccine, or a positive fecal culture of Listeria at screening
2. Currently have or have history of certain study-specified heart, liver, kidney, lung, neurological, immune or other medical conditions
3. Allergy to penicillin or yeast or other component of the study drug product (e.g., glycerol)
4. Clinical metabolic or laboratory abnormalities defined as Grade 3 or 4 of the National Cancer Institute's (NCI's) Common Terminology Criteria for Adverse Events (CTCAE), version 3.0
5. Artificial (prosthetic) joint or other artificial implant or devices that cannot be easily removed
6. Certain types of blood transfusions within 14 days prior to receiving study drug or a condition requiring regular blood transfusions more than twice per month
7. Taking the following medications:

   * Anti-coagulation medications
   * Systemically active steroids for more than 2 days within 28 days prior to receiving study drug
   * More than 325 mg per day of aspirin
   * More than 2 g per day of acetaminophen
   * Systemic antibiotics within 14 days prior to receiving study drug
   * Another investigational product within 28 days prior to receiving study drug
8. Major surgery or significant traumatic injury (or unhealed surgical wounds) occurring within 28 days prior to receiving study drug, or planned surgery requiring general anesthesia
9. Infection with HIV, hepatitis B or C, or HTLV-1 (human t-lymphotropic virus type 1) at screening
10. Pregnant or lactating, or close contact with pregnant women or newborn babies
11. Conditions, including alcohol or drug dependence, intercurrent illness, or lack of sufficient peripheral venous access, that would affect the patient's ability to comply with study visits and procedures

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2007-12; Primary Completion 2009-02 (Actual); Study Completion 2009-02 (Actual)

PRIMARY OUTCOMES:
Dose-limiting toxicities related to the investigational agent | 28 days after first dose

CONTACTS AND LOCATIONS:
Overall Officials: Dung Thai, Study Director — Anza Therapeutics, Inc.
Locations (4):
- United States (3):
  - The Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins University, Baltimore, Maryland
  - National Cancer Institute, NCI, Bethesda, Maryland
  - University of Pennsylvania Abramson Family Cancer Research Center, Philadelphia, Pennsylvania
- Hadassah Hebrew University Medical Center, Jerusalem, Israel